CLINICAL TRIAL: NCT00638378
Title: A Phase 2, Open-Label Study of INCB018424 Administered Orally to Patients With Androgen Independent Metastatic Prostate Cancer
Brief Title: Study of Ruxolitinib (INCB018424) Administered Orally to Patients With Androgen Independent Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: According to the protocol, the sponsor terminated the study after it was determined that less than 2 of the first 22 patients showed a PSA50 response.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-254
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib (Experimental): Participants received ruxolitinib 25 mg orally twice daily in 12-hour intervals for 21-day cycles for as long as the study medication was tolerated and provided clinical benefit.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 25 mg tablets taken with water twice a day.
  Other Names: INCB018424

SUMMARY:
This is a clinical trial of orally administered Ruxolitinib (INCB018424) in patients whose disease has progressed following 1 prior chemotherapy regimen (not including anti-androgens or ketoconazole) for metastatic, androgen-independent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with radiographically-documented metastatic prostate cancer that has progressed while receiving androgen-suppressive therapy in the form of a bilateral orchiectomy or Gonadotropin-Releasing Hormone (GnRH) agonist (eg, leuprolide, goserelin).
* Patients must demonstrate evidence of progressive disease based on 1 of the following criteria: 1) Progressive measurable disease, or 2) Progressive rise in prostate-specific antigen (PSA) level (2 consecutive rises from a prior reference level), or 3) Development of new lesions on bone scan.
* If receiving a GnRH agonist as primary hormonal therapy, the serum testosterone level must be ≤ 50 ng/mL.
* Must have received and progressed during or following 1 prior chemotherapy regimen for metastatic disease (not including an anti-androgen or ketoconazole); or, must have discontinued prior systemic therapy because of poor tolerance or other adverse effects; or, must have refused chemotherapy treatment. Patients having undergone more than 1 prior chemotherapy regimen may be admitted at the discretion of the sponsor.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Baseline serum PSA level of ≥ 10 ng/mL

Exclusion Criteria:

* Received any anti-cancer medications in the 30 days before receiving their first dose of study medication except for GnRH agonists and bisphosphonates.
* Any unresolved toxicity greater than or equal to Grade 2 from previous anti-cancer therapy, except for stable chronic toxicities not expected to resolve, such as peripheral neurotoxicity.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Highland, California
  - Montebello, California
  - Mountain View, California
  - Galesburg, Illinois
  - Overland Park, Kansas
  - Wichita, Kansas
  - Grand Rapids, Michigan
  - Jefferson City, Missouri
  - Great Falls, Montana
  - Cherry Hill, New Jersey
  - Staten Island, New York
  - Bismarck, North Dakota
  - Bethlehem, Pennsylvania
  - Sumter, South Carolina
  - Lacey, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 22
Completed | 0
Not Completed | 22
Not completed — Death | 2
Not completed — Adverse Event | 1
Not completed — Disease progression | 15
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (7.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Prostate-specific Antigen Response
Description: A prostate-specific antigen (PSA) response was defined as a PSA decline from Baseline of 50% or greater, repeated on 2 occasions at least 4 weeks apart.
Time Frame: Assessed monthly from Baseline until the end of study (up to 8 months)
Population: The Intent-to-treat population, which included all patients enrolled in the study who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 22
participants | 0

2. Secondary Outcome: Time to Progression
Description: The time from first dosing day to the date of disease progression:
  * Progressive measurable disease by RECIST criteria (regardless of bone scan or prostate-specific antigen (PSA) results).
  * Development of unequivocal new lesions on bone scan without clinical suspicion of a "flare" reaction.
  * In patients who responded or had a decreased PSA from Baseline, a rise of 50% from PSA nadir, if the increase is ≥ 5 ng/mL or back to Baseline and confirmed by a 2nd value.
  * In patients with no decrease in PSA from Baseline, a 25% rise over Baseline and ≥ 5 ng/mL confirmed by a 2nd value.
Time Frame: From Baseline until the end of study (up to 8 months).
Population: According to the protocol, the sponsor decided to close the study after it was determined that less than 2 of the first 22 patients showed a PSA50 response. Given that all patients discontinued the study due to lack of efficacy, the secondary endpoint of median time to progression was not assessed.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: A treatment-related AE was defined as an event with a definite, probable, or possible causality to study medication. A serious AE is an event resulting in death, hospitalization, persistent or significant disability/incapacity, or is life threatening, a congenital anomaly/birth defect or requires medical or surgical intervention to prevent 1 of the outcomes above. The intensity of an AE was graded according to the National Cancer Institute common terminology criteria for adverse events (NCI-CTCAE) version 3.0: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (life-threatening).
Time Frame: From Baseline through to the end of study (up to 8 months)
Population: The Safety population included all enrolled patients who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 22
Participants
  Any adverse event | 22
  Treatment-related adverse event | 16
  Serious adverse event | 9
  Grade 3 or 4 adverse event | 13
  Discontinued study medication due to adverse event | 4
  Discontinued study due to adverse events | 1

4. Secondary Outcome: Number of Participants With a Complete Response or Partial Response
Description: Complete Response (CR) and Partial Response (PR) defined by the Response Evaluation Criteria in Solid Tumor (RECIST) criteria. CR: Disappearance of all target and nontarget lesions. PR: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter, or persistence of 1 or more nontarget lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: From Baseline through the end of study (up to 8 months)
Population: According to the protocol, the sponsor decided to close the study after it was determined that less than 2 of the first 22 patients showed a PSA50 response. Given that all patients discontinued the study due to lack of efficacy, the secondary endpoint of tumor response rate was not assessed.
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ruxolitinib
Serious Adverse Events (participants affected / at risk) | 9/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=22)
Anaemia (Blood and lymphatic system disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=22)
Anaemia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 9
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 3
Chills (General disorders) | 2
Oedema (General disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Blood lactate dehydrogenase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 2
Weight decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study; provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.